CLINICAL TRIAL: NCT01170598
Title: A Pilot Exercise RCT for Acute Myeloid Leukaemia (AML) Patients Undergoing Induction Chemotherapy: Pre-randomization Phase
Brief Title: Acute Myeloid Leukaemia (AML) Patients Undergoing Induction Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Responsible Party: Principal Investigator, Shabbir Alibhai, Staff Physician and Scientist, Toronto Rehabilitation Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AML002
Record Dates: First submitted 2010-07-21; First posted 2010-07-27 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; AML; chemotherapy; exercise; quality of life; cancer-related fatigue; elderly; physical fitness; muscular strength; Feasibility; Efficacy; Safety
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — After obtaining daily medical clearance, patients will be approached 4-5 days per week to perform 30-45 minutes of supervised exercise with a Canadian Society for Exercise Physiology (CSEP) - Certified Exercise Physiologist. All exercise sessions will be as tolerated, based on patient symptoms.
  Other Names: Mixed-modality exercise; Resistance exercise training; Aerobic exercise training

SUMMARY:
Fatigue, reduced quality of life and declines in physical function are common in patients undergoing chemotherapy for acute myeloid leukaemia (AML). Studies in other cancer patients undergoing treatment have shown that exercise improves these symptoms, but there are limited studies in AML. This study of a hospital-based exercise program will help determine if exercise is both feasible and helpful in improving symptoms among for AML patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Background: Acute myeloid leukaemia (AML) is a life-threatening haematological malignancy. Initial treatment with induction chemotherapy requires 4-5 weeks of hospitalization, with a risk of physical deconditioning, declines in quality of life (QOL), and significant fatigue. Four pilot exercise studies have demonstrated improved fitness, strength, QOL, and fatigue in patients undergoing induction, but are limited by small sample sizes, recruitment of mostly younger adults, inconsistent endpoints, and design issues. Prior to conducting a large multi-centre randomized controlled trial (RCT), important pilot work first needs to be done to demonstrate feasibility of a randomized trial of an exercise program in AML patients undergoing induction chemotherapy; to ensure safety; and to provide effect estimates of the intervention on fitness and QOL/fatigue endpoints.

Objectives: Primary objectives are: (1) to determine feasibility of recruitment and retention of adult AML patients to a randomized trial of supervised exercise and ability of patients to perform an exercise intervention in hospital; (2) to provide estimates of the effect of exercise on fitness parameters. Secondary objectives are: (1) to determine effects of exercise on QOL and fatigue; (2) to understand the impact of exercise on AML treatment tolerability; (3) to examine safety of the exercise intervention. Methods: Thirty-five patients age 18 or older with newly diagnosed or relapsed AML who are undergoing induction chemotherapy will be recruited at Princess Margaret Hospital. Participants will perform 30-45 minutes of supervised aerobic and resistance exercises 4-5 days per week. Primary outcomes are recruitment rate, exercise adherence rate, and impact on fitness measures (peak aerobic capacity (VO2peak), grip strength, leg strength, 6-minute walk test). QOL will be measured with the European Organization for the Research and Treatment of Cancer (EORTC) core 30-item questionnaire (QLQ-C30). Fatigue will be measured using the Functional Assessment of Cancer Therapy fatigue subscale (FACT-Fatigue). Treatment tolerability outcomes include length of stay, intensive care unit admission, and the development of sepsis. Outcomes over time will be assessed using mixed effects regression models.

Significance: Exercise is a promising intervention for improving fitness, QOL and treatment tolerability in AML patients undergoing induction chemotherapy. This pilot RCT will establish feasibility and safety, as well as provide efficacy estimates that will be vital to the design and conduct of a definitive multi-centre RCT of exercise in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* newly diagnosed AML, or relapsed AML after having been in complete remission for at least 6 months
* initiating induction chemotherapy
* ambulatory without need for human assistance
* has consented to study
* is medically cleared for participation by attending physician

Exclusion Criteria:

* has another active malignancy
* has life expectancy < 1 month, physician determined
* has significant comorbidity
* has uncontrolled pain
* has haemodynamic instability
* lacks fluency in reading and writing English and there is no translator available for each visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir MH Alibhai, MD, MSc, Principal Investigator — University Health Network, Toronto Rehab Institute
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Alibhai SM, O'Neill S, Fisher-Schlombs K, Breunis H, Brandwein JM, Timilshina N, Tomlinson GA, Klepin HD, Culos-Reed SN. A clinical trial of supervised exercise for adult inpatients with acute myeloid leukemia (AML) undergoing induction chemotherapy. Leuk Res. 2012 Oct;36(10):1255-61. doi: 10.1016/j.leukres.2012.05.016. Epub 2012 Jun 21. PMID 22726923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-randomized phase II study recruited patients between June 2010 and February 2011. All participants were recruited from Princess Margaret Hospital (PMH) in Toronto, Canada.
Groups:
- Exercise: All study participants were part of the exercise group as this was a non-randomized study. Participants were approached 4-5 times per week to participate in supervised, individualized exercise sessions that incorporated a combination of aerobic, resistance and flexibility exercises. Exercise was light to moderate in intensity and each exercise session was 30-45 minutes in length.
Period: Overall Study
Arm/Group | Exercise
Started | 35
Completed | 29
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Death | 3
Not completed — Lost to Follow-up | 1
Not completed — Refused | 1

BASELINE CHARACTERISTICS:
Arm/Group | Exercise
Number analyzed (Participants) | 35
Age, Customized [Number; unit: years]
  <60 years | 18
  >=60 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Peak Aerobic Capacity (VO2peak)
Description: The modified Bruce protocol is a walking-based treadmill test used to assess peak aerobic capacity. As the test progresses the intensity of each 3-minute work load increases. The test concludes when the participant reaches his maximal heart rate or volitional fatigue. The value attained on this test is measured in metabolic equivalents (METS). METS are a measure of exercise intensity and reflect the physical demands of an activity. In this context, a higher value achieved on the treadmill test (in METS) indicates work at a higher intensity and therefore a higher aerobic capacity.
Time Frame: Baseline, Post-induction (weeks 4-6)
Measure: Mean (Standard Deviation); unit: metabolic equivalent (METS)
Arm/Group | Exercise
Number analyzed (Participants) | 35
metabolic equivalent (METS)
  Baseline | 6.9 (1.8)
  Post-induction (weeks 4-6) | 7.4 (1.7)

2. Primary Outcome: 6-minute Walk Test
Description: Measure of functional endurance assessed by the walking distance covered in a 6-minute period. Participants walk a pre-established course for a total of 6 minutes. The distance covered in that time is recorded as the 6-minute walk test score.
Time Frame: Baseline, Post-induction (4-6 weeks)
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Exercise
Number analyzed (Participants) | 35
feet
  Baseline | 962.5 (286.3)
  Post-induction (weeks 4-6) | 1176.2 (360.6)

3. Primary Outcome: Timed 10-chair Stands
Description: Measure of lower-body strength completed by standing from a seated position 10 times as quickly as possible.
Time Frame: Baseline, Post-induction (weeks 4-6)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Exercise
Number analyzed (Participants) | 35
seconds
  Baseline | 33.0 (26.0)
  Post-induction (weeks 4-6) | 31.1 (11.2)

4. Primary Outcome: Grip Strength
Description: Measure of upper-body strength using a Jamar hand dynamometer. Participants were asked to hold and squeeze (the dynamometer) with maximal force. Three trials were completed with each hand, alternating between the right and left to minimize fatigue. The highest recorded value of the dominant hand was used in the analysis.
Time Frame: Baseline, Post-induction (weeks 4-6)
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Exercise
Number analyzed (Participants) | 35
kilograms
  Baseline | 23.9 (11.0)
  Post-induction (weeks 4-6) | 21.6 (11.0)

5. Secondary Outcome: Global Quality of Life
Description: Global quality of life (QOL) will be measured by the European Organization for the Research and Treatment of Cancer (EORTC) core 30-item questionnaire (QLQ-C30). The EORTC QLQ-C30 is a widely used, self-reported, psychometrically sound cancer QOL instrument. QOL scores derived from this questionnaire range from 0-100 with a higher score reflecting a higher QOL.
Time Frame: Baseline, Post-induction (weeks 4-6)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise
Number analyzed (Participants) | 34
units on a scale
  Baseline | 45.1 (26.6)
  Post-induction (weeks 4-6) | 51.4 (21.4)

6. Secondary Outcome: Fatigue
Description: Fatigue will be assessed using the Functional Assessment of Cancer Therapy fatigue subscale (FACT-Fatigue). The FACT-Fatigue consists of 13 questions and has excellent psychometric characteristics. Fatigue scores derived from this questionnaire range from 0-52 with a higher score reflecting lower fatigue.
Time Frame: Baseline, Post-induction (weeks 4-6)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise
Number analyzed (Participants) | 34
units on a scale
  Baseline | 31.5 (13.1)
  Post-induction (weeks 4-6) | 33.9 (11.7)

7. Secondary Outcome: Length of Stay
Description: Length of stay (date of admission to hospital to date of discharge).
Time Frame: Post-induction (weeks 4-6)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Exercise
Number analyzed (Participants) | 34
days | 37.2 (10.6)

8. Secondary Outcome: Intensive Care Unit (ICU) Admission
Description: Intensive care unit (ICU) admission (percentage of participants admitted to ICU during induction chemotherapy course).
Time Frame: Post-induction (weeks 4-6)
Measure: Number; unit: percentage of participants
Arm/Group | Exercise
Number analyzed (Participants) | 34
percentage of participants | 11.5

9. Secondary Outcome: Development of Sepsis
Description: Development of sepsis (percentage of participants who developed sepsis during induction chemotherapy course).
Time Frame: Post-induction (weeks 4-6)
Measure: Number; unit: percentage of participants
Arm/Group | Exercise
Number analyzed (Participants) | 34
percentage of participants | 26.5

10. Primary Outcome: Recruitment Rate
Description: Ratio of patients who consented to participate out of all eligible patients expressed as a percentage (eligible patients who consented to participation/eligible patients who declined participation).
Time Frame: Baseline
Population: For this outcome measure we analyzed 52 participants (rather than 35). Fifty-two participants met the study eligibility criteria. Thirty-five out of 52 consented to participate which is how we derived our recruitment rate of 67% (35/52).
Measure: Number; unit: percentage of patients
Arm/Group | Exercise
Number analyzed (Participants) | 52
percentage of patients | 67

11. Primary Outcome: Retention
Description: Percentage of participants who remained in the study (did not withdraw voluntarily).
Time Frame: Baseline, Post-induction (weeks 4-6)
Measure: Number; unit: percentage of participants
Arm/Group | Exercise
Number analyzed (Participants) | 35
percentage of participants | 97

12. Primary Outcome: Program Adherence.
Description: Adherence to supervised exercise program assessed as a percentage of exercise sessions completed(number of days of supervised exercise performed/the number of days that patients were approached to participate).
Time Frame: Baseline, Post-induction (weeks 4-6)
Measure: Number; unit: percentage of exercise days completed
Arm/Group | Exercise
Number analyzed (Participants) | 34
percentage of exercise days completed | 45.8

ADVERSE EVENTS:
Time Frame: Adverse event data were captured over the course of the intervention (9 months).
Description: Any adverse events were captured using the National Cancer Institute: Cancer Therapy Evaluation Program Common Terminology Criteria version 3.0.
Arm/Group | Exercise
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 1/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise (N=35)
Possible grade II musculoskeletal event (Musculoskeletal and connective tissue disorders) | 1 (1) — In over 600 patient-days of observation, one possible grade II musculoskeletal event occurred (neck/back pain limiting function for 24 hours). No other adverse events or safety concerns were reported.

LIMITATIONS AND CAVEATS:
Although as per study design, limitations include the lack of a control group due to non-randomization, a small sample size and lack of generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes